CLINICAL TRIAL: NCT04615858
Title: Genepro Generation 3 Bioavailability Compared to Whey Protein (12g Genepro vs 30g Whey)
Brief Title: Genepro Generation 3 Protein Bioavailability Compared to Whey Protein
Acronym: Gen3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Musclegen Research, Inc. (Other)
Collaborators: WakeMed Bariatric Surgery & Weight Loss Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Genepro Gen3; 033300391 (Other: US DOD); Patent Pending (Other: USPTO)
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Absorption; Disorder, Protein; Protein Malabsorption; Protein Intolerance
Keywords: protein; absorption
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Masking Description: Active Comparator: Genepro Gen2 Protein 11g Serving of Genepro Gen3 Protein daily will be used in each subject. Intervention: Bi-Weekly blood draws will determine the effect on blood protein levels.
  Active Comparator: Whey Protein Isolate 30g Serving of Whey Protein will be used daily in each subject. Intervention:Bi-Weekly blood draws will determine the effect on blood protein levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genepro Generation 3 (Active Comparator): 1 scoop, 11g, Genepro Generation 3 Protein daily will be used by Group A (20 participants) 10 male, 10 female participants 6 months post bariatric surgery.
  Interventions: Dietary Supplement: Genepro Generation 3 Protein
- Whey Protein (Active Comparator): 1 scoop, 30g, Whey Protein daily will be used by Group B (20 participants) 10 male, 10 female participants 6 months post bariatric surgery.
  Interventions: Dietary Supplement: Whey Protein

INTERVENTIONS:
Dietary Supplement: Genepro Generation 3 Protein — Generation 3 Genepro Protein. Micronized protein. Zero lactose. No gluten. All Natural. No flavor. No Sugar. FODMAP Certified protein. 11g in weight, scoop.
  Arms: Genepro Generation 3
Dietary Supplement: Whey Protein — Nutrition industries number 1 selling whey protein powder. No flavor. Gluten Free. 30g scoop.
  Arms: Whey Protein

SUMMARY:
Objective of Clinical Trial: To test, in a blinded study the bioavailability of Genepro Generation 3 (GEN3) Protein as compared to whey protein. This study is intended to show the equivalent value of Genepro Gen3 as compared to whey protein (1scoop (12g) Genepro Generation 3 (GEN3) compared to 30g serving of whey protein). Total Serum Protein levels will be tested every other week to evaluate blood protein levels in each participant

DETAILED DESCRIPTION:
Detailed Description:

Condition or Disease: Analysis, Event History. Absorption; Disorder, protein

Objective of Clinical Trial: To test, in a blinded study the bioavailability of Genepro Generation 3 (GEN3) Protein as compared to whey protein. This study is intended to show the equivalent value of Genepro Gen3 as compared to whey protein (1scoop (12g) Genepro Generation 3 (GEN3) compared to 30g serving of whey protein). Total Serum Protein levels will be tested every other week to evaluate blood protein levels in each participant.

Parameters: This study encompasses a 6-week program that follows 40 gastric bypass patients that have undergone weight loss surgery. We will establish a baseline blood analysis prior to the start of the study and subsequently we will take bi-weekly blood work to chart and register the findings (weeks 2, 4 and 6). For this study we will only be doing the bi-weekly analysis on blood protein levels by utilizing Spectrophotometry with total serum protein. The target blood protein range is 6.1-8.7 g/dL this test is administered without fasting.

Participants: 40 Post Op Gastric Bypass patients. 20 men, 20 women. All participants were between the ages of 25-80 years of age. All participants have been post operation from their weight loss surgery for a minimum of 6 months prior to the start of the study and no longer than 8 months at the start of the study. Participants will be randomly selected, blindly, by the study sponsor. The selection will utilize participants files with names and ethnicity removed. Selection will be randomized into Group A and Group B. One group will be assigned Genepro while the other group will be assigned a leading whey protein powder. Participants will be assigned a Identification Code/Number for the duration of the study. Results will be posted using this identification number as well as stating the age and gender of the participant. Participant names will be held in confidence. Participants must maintain a daily log that will be shared with study investigators. This log will contain daily lists of food and beverage consumed as well as personal thoughts on taste and ease of use of protein supplements as well as a daily synopsis of overall general emotional and physical feelings.

Participant Compensation: Three (3) thirty serving units of Genepro Generation 3 at the conclusion of the study.

Gathering Results: 40 subjects will receive Genepro Generation 3 protein (12g serving) for one week prior to the study as well as all 6 weeks of the study. In conjunction the other group of 20 subjects will receive 30g whey protein for one week prior to the study as well as all 6 weeks of the study. Bi-Weekly blood analysis will determine blood protein levels. Blood draws are to be conducted at a WakeMed facility (Cary, NC or Raleigh, NC - determined by the proximity to the patient for their convenience). Results will be submitted for review and entry from WakeMed to the sponsor oversight POC every 2 weeks. To ensure proper transfer of data, WakeMed will keep and store all lab reports/results for a minimum of 2 years after the conclusion of the study. Soft copies will be inserted into a virtual storage center to be maintained and accessible by both, the sponsor as well as the medical partners.

Diet: Diet guidelines limit the calories you consume while providing you with balanced meals to help prevent nutritional deficiencies and preserve your muscle tissue. Each patient tolerates suggested foods differently. Daily calories should be between 600 to 700 for the duration of this study. Each subject is to follow a diet low in calories, fats and sweets. The goal for each subject is to consume a minimum of 65 to 75 grams of protein a day. High protein foods include eggs, meats, fish, seafood, tuna, poultry, tofu, milk, soy, cottage cheese, and yogurt. 30g of each daily intake of protein will be provided by a powdered protein supplement. 20 subjects will utilize a 30g serving of whey protein for 1 week prior to the study as well as 6 weeks of the study. The other group of 20 subjects will use a single serving (12g) of Genepro Gen3 Protein over the same duration.

Subject were given the following eating guidelines:

* Eat slowly and chew small bites of food thoroughly.
* Avoid rice, bread, raw vegetables, fresh fruits, and meats that are not easily chewed such as pork and steak. Ground meats are usually better tolerated.
* With soft and solid foods, take only three bites at one sitting, then wait a minimum of 20 minutes before eating more.
* Eat balanced meals with small portions.
* Avoid the use of drinking straws and carbonated beverages, chewing gum and ice because they can introduce too much air into your pouch and cause discomfort.
* Avoid sugar, sugar-containing foods and beverages, concentrated sweets, and fruit juices Alcoholic beverages will have a more profound effect and should be avoided or consumed with caution.

Storage and Distribution of Protein Powder: WakeMed Clinical Oversight Manager and Principal Investigator, Marina Maddaloni, will be provided with a lockable storage container to be positioned in her personal office. WakeMed will be provided white and black containers. One color will house either Genepro or regular Whey protein. WakeMed will not have knowledge of which color container holds which protein powder to ensure that the distribution to participants is totally blinded. Participants will be given enough protein supplementation, either regular whey or Genepro Generation 3 protein, to last the duration of the study.

Peer Reviewer 1: Dr. Brian M. Parks Peer Reviewer 2: Zac Cain Non-Peer Review: Dr. Jon Bruce

ELIGIBILITY:
INCLUSION CRITERIA:

* Participants will be solicited to volunteer through WakeMed Bariatric Surgery Center (current patients)
* All participants must have normal blood protein levels prior to the study
* All participants must be six months post op (bariatric surgery)
* All participants must avoid any other protein supplementation during the trial period
* All participants are required to maintain a daily nutrition log
* All participants must have no milk/dairy allergies
* Age Eligibility: 25 years to 80 years (Adult)
* Sexes Eligibility for Study: ALL
* Only Accepts Healthy Volunteers

EXCLUSION CRITERIA:

* No candidates with prior digestive distress disorders (IBS, Crones, etc.)
* Participants with any negative GI score, they will be excluded from the study
* Participants with abnormal blood protein levels at the time of study
* Unhealthy Volunteers
* Volunteers with compromised immune systems
* Volunteers younger than 25 years of age
* Volunteers older than 80 years of age
* Allergies to milk or lactose

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-01-26 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood Protein Levels | 6 weeks
  Each participant in each group will have blood protein levels checked via blood draw at a WakeMed facility (based on participants geographic location). The target blood protein range is 6.1-8.7 g/dL this test is administered without fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Maddaloni, Study Chair — WakeMed Bariatric Surgery Center; Zac Cain, Study Chair — Genepro Protein, Inc.; Brian Parks, PHD, Study Director — Genepro Protein, Inc.; John Bruce, MD, Principal Investigator — WakeMed Bariatric Surgery Center; LaMonica Daniel, Study Chair — WakeMed Health & Hospitals
Locations (2):
- United States (2):
  - WakeMed Bariatric Surgery Center, Cary, North Carolina
  - WakeMed, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No